CLINICAL TRIAL: NCT03178734
Title: Foley Catheter vs a Self-contained Valved Urinary Catheter for Patients Who Are Being Discharged Home With a Catheter After Urogynecologic Procedures
Brief Title: Foley Catheter vs a Self-contained Valved Urinary Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: charbel salamon (Other)
Responsible Party: Sponsor-Investigator, charbel salamon, Charbel Salamon, MD, MS, FACOG, Atlantic Health System
Organization: Atlantic Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 908398
Record Dates: First submitted 2017-05-11; First posted 2017-06-07 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Catheter-Related Infections; Urinary Tract Infections; Urogynecologic Surgery
MeSH Terms: conditions — Catheter-Related Infections; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: This study aim is to compare UTI rates and patient satisfaction associated with indwelling Foley catheter vs a valved catheter in patients who are being discharged home with a catheter after urogynecologic proecures via a Randomized Clinical Trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Indwelling Foley Catheter (Other): These patients will have a traditional foley catheter with attached drainage bag (Indwelling Foley Catheter).
  Interventions: Device: Foley Catheter vs Self-Contained Valved Catheter
- Self-Contained Valved Catheter (Other): These patients will have a BARD Flip Flo Catheter Valve attached to the original foley catheter (Self-Contained Valved Catheter).
  Interventions: Device: Foley Catheter vs Self-Contained Valved Catheter

INTERVENTIONS:
Device: Foley Catheter vs Self-Contained Valved Catheter — This study aims to compare UTI rates and patient satisfaction between an indwelling Foley catheter group (established SOC); and a relatively (FDA-approved) new valved addition to the Foley catheter which requires no drainage bag.

SUMMARY:
The purpose of this study is to compare UTI rates and patient satisfaction associated with indwelling Foley catheter verses a valved catheter in patients who are being discharged home with a catheter after urogynecologic procedures via a Randomized Clinical Trial.

DETAILED DESCRIPTION:
The purpose of this study is to compare UTI rates and patient satisfaction associated with indwelling Foley catheter verses a valved catheter in patients who are being discharged home with a catheter after urogynecologic procedures via a Randomized Clinical Trial. Total number of participants will be 100. Inclusion criteria is all patients undergoing pelvic reconstructive surgery/anti-incontinence procedures who are planned to be discharged home with a catheter. Exclusion criteria is intra-operative bladder injury during index surgery; intra-operative complication requiring continuous bladder drainage; and/or dementia/altered cognitive function.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing pelvic reconstructive surgery/anti-incontinence procedures who are planned to be discharged home with a catheter.

Exclusion Criteria:

* Intra-operative bladder injury during index surgery
* Intra-operative complication requiring continuous bladder drainage
* Dementia / altered cognitive function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of urinary tract infections | Up to 4 weeks after surgery
  Number of urine cultures positive for infection (taken at voiding trial visit and post-operative visit).

SECONDARY OUTCOMES:
Patient satisfaction | Up to 5 days after surgery
  Foley satisfaction questionnaire will be collected at post-operative voiding trial office visit.
Number of days until spontaneous void/Number of calls for device-related issues | Up to 4 weeks after surgery
  Number of days until spontaneous void and number of call for device-related issues.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel G Salamon, MD, MS, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Urogynecology Associates, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246